CLINICAL TRIAL: NCT04534842
Title: An Open-label Study of the Efficacy and Safety of SYNB1618 and SYNB1934 in Patients With Phenylketonuria (SynPheny-1)
Brief Title: Efficacy and Safety of SYNB1618 and SYNB1934 in Adult Patients With Phenylketonuria
Acronym: SynPheny-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Synlogic (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYNB1618-CP-003
Record Dates: First submitted 2020-08-24; First posted 2020-09-01 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Phenylketonuria
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SYNB1618 (Experimental): Dose ramp of SYNB1618
  Interventions: Drug: SYNB1618
- SYNB1934 (Experimental): Dose ramp of SYNB1934
  Interventions: Drug: SYNB1934

INTERVENTIONS:
Drug: SYNB1618 — 15-day dose-ramp regimen (4 dose levels) of orally administered SYNB1618
  Arms: SYNB1618
Drug: SYNB1934 — 15-day dose-ramp regimen (4 dose levels) of orally administered SYNB1934
  Arms: SYNB1934

SUMMARY:
This Phase 2 study in patients with phenylketonuria (PKU) will be an open-label, dual-arm study of either a SYNB1618 or SYNB1934 dose-ramp regimen. All evaluations and assessments throughout this study may be conducted either at the clinical site or by a home healthcare professional at an alternative location (e.g., patient's home, hotel).

DETAILED DESCRIPTION:
This is an open-label, dual-arm Phase 2 study; all participating PKU patients will receive active study drug, SYNB1618 or SYNB1934. This study is evaluating a dose-ramp regimen consisting of 4 dose levels of SYNB1618 or SYNB1934 over 15 days of treatment.

This study has been designed with the flexibility of being able to be conducted either at the clinical site or by a home healthcare professional at an alternative location (e.g., patient's home, hotel).

Patients will be screened for eligibility and complete a customized diet run-in period prior to starting the 15-day dose ramp ('treatment period'). During the treatment period patients will be required to adhere to the same customized diet menus as in the diet run-in period.

The efficacy of SYNB1618 SYNB1934 will be assessed in this study by measuring the reduction of the area under the curve (AUC) for plasma D5-phenylalanine (D5-Phe) as well as the reduction of plasma Phe levels.

Safety will be monitored by documentation of adverse events (AEs), clinical laboratory measurements, vital signs, and physical examinations.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Able and willing to voluntarily complete the informed consent process.
3. Diagnosis of classic PKU based on medical history as assessed by the investigator (e.g., Phe concentration of >1200 µmol/L at any time, low dietary Phe tolerance, or genetic diagnosis).
4. Blood Phe ≥ 600 µmol/L at Screening.
5. Stable diet including stable medical formula regimen (if used) for at least 1 month prior to Screening.
6. Available for and agree to all study procedures, including urine and blood collection, adherence to diet control, follow-up visits, and IMP ingestion compliance.
7. Male patients who are sexually abstinent or surgically sterilized (vasectomy), or those who are sexually active with a female partner(s) and agree to use an effective method of contraception (such as condom with spermicide) combined with an acceptable method of contraception for their non-pregnant female partner(s) (as defined in Inclusion Criterion #8 below) after informed consent, throughout the study, and for a minimum of 3 months after the last dose of IMP, and who do not intend to donate sperm in the period from Screening until 3 months following administration of the IMP.
8. Female patients who meet one of the following criteria:

   1. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test (human chorionic gonadotropin) at Screening and a negative urine pregnancy test at Baseline prior to the start of IMP and must agree to use acceptable method(s) of contraception, combined with an acceptable method of contraception for their male partner(s) (as defined in Inclusion Criterion #7 above) after informed consent, throughout the study, and for a minimum of 3 months after the last dose of IMP. Acceptable methods of contraception include hormonal contraception, hormonal or non-hormonal intrauterine device, bilateral tubal occlusion, complete abstinence, vasectomized partner with documented azoospermia 3 months after procedure, diaphragm with spermicide, cervical cap with spermicide, vaginal sponge with spermicide, or male or female condom with or without spermicide.
   2. Premenopausal woman with one of the following:

   i. Documented hysterectomy, ii. Documented bilateral salpingectomy, iii. Documented bilateral oophorectomy, iv. Documented tubal ligation/occlusion, v. Sexual abstinence is preferred or usual lifestyle of the patient c. Postmenopausal women (12 months or more amenorrhea verified by follicle stimulating hormone [FSH] assessment and over 45 years of age, in the absence of other biological or physiological causes).
9. Screening laboratory evaluations (e.g., chemistry panel, complete blood count [CBC] with differential, urinalysis, creatinine clearance, CRP) within normal limits or judged to be not clinically significant by the investigator.

Exclusion Criteria:

1. Currently taking Palynziq® (pegvaliase-pqpz) (within 1 month of Screening).
2. Inflammatory or irritable bowel disorder of any grade.
3. History of or current immunodeficiency disorder.
4. Intolerance of or allergic reaction to E. coli Nissle or any of the ingredients in SYNB1618 formulation.
5. Any condition (e.g., celiac disease, gastrectomy, bypass surgery, ileostomy) or receiving prescription medication or an over-the-counter product that may possibly affect absorption of medications or nutrients.
6. Currently taking or plans to take any type of systemic (e.g., oral or intravenous) antibiotic within 28 days prior to the first dose of IMP through final safety assessment, including planned surgery, hospitalizations, dental procedures, or interventional studies that are expected to require antibiotics. Exception: topical antibiotics are allowed.
7. Within the 3 months prior to anticipated first dose, major surgery (an operation upon an organ within the cranium, chest, abdomen, or pelvic cavity) or inpatient hospital stay.
8. Dependence on alcohol or drugs of abuse.
9. Administration or ingestion of an investigational drug within the 30 days or 5 half-lives before Screening, whichever is longer, or cell/gene therapy prior to the Screening visit, or current enrollment in an investigational drug study.
10. Acute or chronic medical, surgical, psychiatric, or social condition or laboratory abnormality that may increase patient risk associated with study participation, compromise adherence to study procedures and requirements, or may confound interpretation of study safety or PD results and, in the judgment of the investigator, would make the patient inappropriate for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in labeled Phe (D5-Phe) in plasma | Day 14
  The primary efficacy outcome will be assessed by measuring change from baseline in plasma D5-Phe AUC over 24 hours after D5-Phe administration

SECONDARY OUTCOMES:
Changes from baseline in fasting levels of plasma Phe | Day 14
  The secondary efficacy outcome will be assessed by measuring fasting levels of plasma Phe as compared to baseline
Incidence of Treatment-Emergent Adverse Events | Day 43
  Will be measured by assessing nature and frequency of AEs

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Children's Hospital Colorado, Aurora, Colorado
  - Excel Medical Clinical Trials, LLC, Boca Raton, Florida
  - University of Florida College of Medicine, Gainesville, Florida
  - Washington University in St Louis, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Health Science Center at Houston, Houston, Texas
  - PRA Health Sciences, Salt Lake City, Utah
  - University Hospital Adult Services, Salt Lake City, Utah

REFERENCES:
- [Derived] Vockley J, Sondheimer N, Puurunen M, Diaz GA, Ginevic I, Grange DK, Harding C, Northrup H, Phillips JA 3rd, Searle S, Thomas JA, Zori R, Denney WS, Ernst SL, Humphreys K, McWhorter N, Kurtz C, Brennan AM. Efficacy and safety of a synthetic biotic for treatment of phenylketonuria: a phase 2 clinical trial. Nat Metab. 2023 Oct;5(10):1685-1690. doi: 10.1038/s42255-023-00897-6. Epub 2023 Sep 28. PMID 37770764